CLINICAL TRIAL: NCT02170441
Title: Global Consortium for Drug-resistant Tuberculosis Diagnostics
Acronym: GCDD
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Antonino Catanzaro, Professor, University of California, San Diego
Other Study IDs: 09-0099; U01AI082229 (NIH)
Record Dates: First submitted 2014-06-12; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Tuberculosis; Tuberculosis, Multidrug-Resistant
Keywords: Tuberculosis; Multi-drug resistant tuberculosis; Extensively drug-resistant tuberculosis; Drug-resistant tuberculosis; Mycobacterial Growth Indicator Tube Drug Susceptibility Test; Line Probe Assay; Microscopic Observation Drug Susceptibility Assay; Pyrosequencing
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cultured isolates, processed sputum, extracted DNA (crude lysate from sputum)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients at risk for drug-resistant TB: No intervention

SUMMARY:
The goal of this study is to evaluate time to diagnosis for three assays (line probe, pyrosequencing, and Microscopic Observation Drug Susceptibility Assay [MODS]) to detect resistance to first and second-line anti-tuberculosis (TB) drugs in Mycobacterium tuberculosis (Mtb) strains in 7 days or less, allowing for rapid diagnosis of extensively drug-resistant TB (XDR-TB).

DETAILED DESCRIPTION:
The goals of this study are to test, fine tune, and compare three tests (line probe, pyrosequencing, MODS assays) to rapidly detect Mycobacterium tuberculosis (Mtb) strains that are resistant to first and second-line anti-tuberculosis (TB) drugs allowing for rapid diagnosis of Extensively Drug-Resistant Tuberculosis (XDR-TB).

Primary Specific Aims

Aim 1: To reduce the average XDR-TB detection time from months to a week.

Aim 2: To determine agreement between rapid tests and standard drug susceptibility testing (DST) results.

Aim 3: To identify the genetic basis of discordant results from Aim 2.

Aim 4: To characterize genotypic, phenotypic and epidemiological features, as well as geographical relationships, of XDR-TB strains compared to other drug-resistant and susceptible strains.

Secondary Aims Aim 1: Cost-effectiveness study. The costs associated with rapid-test implementation will be compared with the performance of the new tests to rapidly and accurately detect drug resistance and XDR-TB.

Aim 2: To determine the predictive value of resistance-associated mutations in determining sputum culture conversion.

The investigators hypothesize that analysis of the genotypic basis of anti-TB drug resistance will allow for the development of improved rapid molecular drug susceptibility tests that will detect resistance to fluoroquinolones and injectable anti-TB drugs and reduce the current XDR-TB diagnosis time of up to three months to less than seven days.

ELIGIBILITY:
Inclusion Criteria:

* At least 5 years of age
* Known to be acid fast bacilli (AFB) sputum smear-positive, 1+ or greater (within prior 14 days), positive on GeneXpert, or present clinically with high suspicion of active TB and:
* Had previously received >1 month of treatment for a prior TB episode or
* Were failing TB treatment with positive sputum smear or culture after ≥3 months of a standard TB treatment or
* Had had close contact with a known drug-resistant TB case or
* Were newly diagnosed with multi-drug resistant TB (MDR-TB) within the last 30 days or
* Were previously diagnosed with MDR-TB and failed TB treatment with positive sputum smear or culture after ≥3 months of a standard MDR-TB treatment regimen
* Provided informed consent or had ability and willingness of subject or legal guardian/representative to provide informed consent

Exclusion Criteria:

* Institutionalized
* Unable to provide at least 7.5ml sputum (1st and 2nd samples combined)
* Had results from second line DST performed within the last 3 months

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed or previously treated tuberculosis who are at risk for drug-resistant tuberculosis
Sampling Method: Non-Probability Sample
Enrollment: 1128 (Actual)
Dates: Start 2012-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Time to completion of rapid diagnostic assays | Up to 83 weeks
  Time to completion was calculated from date of initial sputum collection to completion of each rapid diagnostic assay. Time frame for analysis of all results was from date of first patient recruited till 21 weeks after last patient recruited (total 83 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Catanzaro, MD, Principal Investigator — University of California, San Diego
Locations (3):
- P.D. Hinduja National Hospital and Medical Research Centre, Mumbai, India
- Phthisiopneumology Institute, Chisinau, Moldova
- Department of Biomedical Sciences, Stellenbosch University, Cape Town, South Africa

REFERENCES:
- [Derived] Groessl EJ, Ganiats TG, Hillery N, Trollip A, Jackson RL, Catanzaro DG, Rodwell TC, Garfein RS, Rodrigues C, Crudu V, Victor TC, Catanzaro A. Cost analysis of rapid diagnostics for drug-resistant tuberculosis. BMC Infect Dis. 2018 Mar 2;18(1):102. doi: 10.1186/s12879-018-3013-0. PMID 29499645
- [Derived] Seifert M, Georghiou SB, Garfein RS, Catanzaro D, Rodwell TC. Impact of Fluoroquinolone Use on Mortality Among a Cohort of Patients With Suspected Drug-Resistant Tuberculosis. Clin Infect Dis. 2017 Sep 1;65(5):772-778. doi: 10.1093/cid/cix422. PMID 28475735
- [Derived] Georghiou SB, Seifert M, Catanzaro DG, Garfein RS, Rodwell TC. Increased Tuberculosis Patient Mortality Associated with Mycobacterium tuberculosis Mutations Conferring Resistance to Second-Line Antituberculous Drugs. J Clin Microbiol. 2017 Jun;55(6):1928-1937. doi: 10.1128/JCM.00152-17. Epub 2017 Apr 12. PMID 28404672
- [Derived] Catanzaro DG, Trollip AP, Seifert M, Georghiou SB, Garfein RS, Rodwell TC, Catanzaro A, Eisenach KD. Evaluation of the microscopic observation drug susceptibility assay for the detection of first- and second-line drug susceptibility for Mycobacterium tuberculosis. Eur Respir J. 2017 Apr 5;49(4):1602215. doi: 10.1183/13993003.02215-2016. Print 2017 Apr. PMID 28381434
- [Derived] Georghiou SB, Seifert M, Lin SY, Catanzaro D, Garfein RS, Jackson RL, Crudu V, Rodrigues C, Victor TC, Catanzaro A, Rodwell TC. Shedding light on the performance of a pyrosequencing assay for drug-resistant tuberculosis diagnosis. BMC Infect Dis. 2016 Aug 31;16(1):458. doi: 10.1186/s12879-016-1781-y. PMID 27576542
- [Derived] Georghiou SB, Seifert M, Catanzaro D, Garfein RS, Valafar F, Crudu V, Rodrigues C, Victor TC, Catanzaro A, Rodwell TC. Frequency and Distribution of Tuberculosis Resistance-Associated Mutations between Mumbai, Moldova, and Eastern Cape. Antimicrob Agents Chemother. 2016 Jun 20;60(7):3994-4004. doi: 10.1128/AAC.00222-16. Print 2016 Jul. PMID 27090176
- [Derived] Hillery N, Groessl EJ, Trollip A, Catanzaro D, Jackson L, Rodwell TC, Garfein RS, Lin SY, Eisenach K, Ganiats TG, Park D, Valafar F, Rodrigues C, Crudu V, Victor TC, Catanzaro A. The Global Consortium for Drug-resistant Tuberculosis Diagnostics (GCDD): design of a multi-site, head-to-head study of three rapid tests to detect extensively drug-resistant tuberculosis. Trials. 2014 Nov 6;15:434. doi: 10.1186/1745-6215-15-434. PMID 25377177
- See also: Related Info — http://gcdd.ucsd.edu